CLINICAL TRIAL: NCT02616991
Title: Contribution of CT Venography for Diagnosing Venous Thromboembolism During Postpartum
Brief Title: Computed Tomography CT Venography During Postpartum Venous Thromboembolism
Acronym: CTVENPOSTPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-002741-64; 2015-A01262-47 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental): computed tomography venography
  Interventions: Procedure: computed tomography venography

INTERVENTIONS:
Procedure: computed tomography venography — systematically performing computed tomography venography in addition to thoracic computed tomography angiography

SUMMARY:
The purpose of this study is to determine whether systematically performing computed tomography (CT) venography (i.e a CT acquisition of the pelvis and of the lower limbs, during the venous phase of opacification) in addition to thoracic CT angiography in women with suspected postpartum pulmonary embolism (PE) results in a gain in venous thromboembolism detection rate.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) remains a leading cause of maternal death during postpartum in developed countries; Thoracic computed tomography angiography (CTA) is the first-line diagnostic test for PE suspicion, but has a 20 to 35% rate of inconclusiveness during pregnancy and postpartum, 2 to 3 times higher than that of the general population. CT venography (CTV) consists in a delayed CT acquisition of the abdomen, pelvis and lower limbs, 3 minutes after starting contrast administration. It can be used for detecting deep venous thrombosis (DVT), the source of emboli in most PEs. The investigators hypothesized most postpartum PEs are due to pelvic vein thrombosis and that detecting such pelvic DVT by performing systematic CTV could increase the overall venous thromboembolism (VTE) detection.

ELIGIBILITY:
Inclusion Criteria:

* Women with clinically suspected pulmonary embolism (PE) during the first 6 weeks postpartum, without any sign of severe PE (shock, hypotension), referred for CT angiography
* Absence of contraindication to iodinated contrast medium injection (Previous allergic reaction to iodinated contrast medium, renal insufficiency with creatine clearance less than 30mL/mn, uncontrolled hyperthyroidism)
* Age > 18 years
* Health insurance
* Possibility to have 3-month follow-up
* Obtention of written informed consent (ability to give consent)

Exclusion Criteria:

* Anticoagulation at therapeutic dosage for another reason than the suspicion of PE for more than 72 hours
* New pregnancy (In case of any doubt after medical history review, βHCG blood test must be realized to ensure patient's pregnancy status)
* Contrast medium extravasation during injection
* CTA or CTV not performed according to the study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-06-04 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Number of detected venous thromboembolism (VTE) based on Computed Tomography Angiography (CTA) plus Computed Tomography Venography (CTV) | one day
  VTE detection rate for readings based on CTA plus CTV as compared to readings based on CTA alone

SECONDARY OUTCOMES:
Radiation doses due to CT venography | 3 months
kappa coefficients assessing inter-readers agreement for CT venography readings | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre REVEL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Guy MEYER, PhD, Study Chair — University of Paris 5 - Rene Descartes
Locations (1):
- Cochin Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revel MP, Chassagnon G, Sanchez O, Ferretti G, Millet I, Rocher L, Maitre S, Lederlin M, Ducou-le-Pointe H, Rousset P, Bennani S, Zins M, Bruneau B, Tissot V, Alison M, Canniff E, Siauve N, Vandeventer S, Le Blanche AF, Planquette B, Tsatsaris V, Coste J. CT venography for the diagnosis of postpartum venous thromboembolism: a prospective multi-center cohort study. Eur Radiol. 2024 Nov;34(11):7419-7428. doi: 10.1007/s00330-024-10791-8. Epub 2024 May 23. PMID 38782788
- [Background] Revel MP, Sanchez O, Dechoux S, Couchon S, Frija G, Cazejust J, Chatellier G, Meyer G. Contribution of indirect computed tomographic venography to the diagnosis of postpartum venous thromboembolism. J Thromb Haemost. 2008 Sep;6(9):1478-81. doi: 10.1111/j.1538-7836.2008.03078.x. Epub 2008 Jul 8. PMID 18627442